CLINICAL TRIAL: NCT05029856
Title: A Randomized, Observer-Blinded, Phase 1/2 Study With an Open-Label Group to Evaluate the Safety and Immunogenicity of SII Vaccine Constructs Based on SARS-CoV-2 Variants in Adults
Brief Title: Evaluation of the Safety and Immunogenicity of SII Vaccine Constructs Based on the SARS-CoV-2 (COVID-19) Variant in Adults
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Study never started
Sponsor: Novavax (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2019nCoV-102
Record Dates: First submitted 2021-08-25; First posted 2021-09-01 (Actual); Last update posted 2022-05-31 (Actual); Status verified 2022-05

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19 | interventions — YY1 Transcription Factor

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- Group A- SII B.1.351 Vaccine / Matrix-M1 Adjuvant (Experimental): 2 doses of 3 μg SII B.1.351 Vaccine+ 50 μg Matrix-M1 adjuvant (co-formulated) . 1 dose each on Days 0 and Day 21.
  Interventions: Biological: SII B.1.351
- Group B- SII B.1.351 Vaccine / Matrix-M1 Adjuvant (Experimental): 2 doses of 5 μg SII B.1.351 Vaccine+ 50 μg Matrix-M1 adjuvant (co-formulated) . 1 dose each on Days 0 and Day 21.
  Interventions: Biological: SII B.1.351
- Group C- SII B.1.351 Vaccine / Matrix-M1 Adjuvant (Experimental): 1 dose of 3 μg SII B.1.351 Vaccine+ 50 μg Matrix-M1 adjuvant (co-formulated) .1 dose on Day 0.
  Interventions: Biological: SII B.1.351
- Group D - SII B.1.351 Vaccine / Matrix-M1 Adjuvant (Experimental): 1 dose of 5 μg SII B.1.351 Vaccine + 50 μg Matrix-M1 adjuvant (co-formulated) .1 dose on Day 0.
  Interventions: Biological: SII B.1.351
- Group E -SII Bivalent Vaccine / Matrix-M1 Adjuvant (Experimental): 2 doses of 6 μg SII Bivalent Vaccine+ 50 μg Matrix-M1 adjuvant (co-formulated) . 1 dose each on Days 0 and Day 21.
  Interventions: Biological: SII Bivalent
- Group F- SII Bivalent Vaccine / Matrix-M1 Adjuvant (Experimental): 2 doses of 10 μg SII Bivalent Vaccine+ 50 μg Matrix-M1 adjuvant (co-formulated) . 1 dose each on Days 0 and Day 21.
  Interventions: Biological: SII Bivalent
- Group G- SII B.1.617.2 Vaccine / Matrix-M1 Adjuvant (Experimental): 2 doses of 5 μg SII B.1.617.2 Vaccine+ 50 μg Matrix-M1 adjuvant (co-formulated) . 1 dose each on Days 0 and Day 21.
  Interventions: Biological: SII B.1.617.2
- Group H- SII B.1.617.2 Vaccine / Matrix-M1 Adjuvant (Experimental): 1 doses of 5 μg SII B.1.617.2 Vaccine+ 50 μg Matrix-M1 adjuvant (co-formulated) . 1 dose on Days 0.
  Interventions: Biological: SII B.1.617.2

INTERVENTIONS:
Biological: SII B.1.351 — Intramuscular (deltoid) injections of 3 μg SII B.1.351 and 50 μg Matrix-M1 Adjuvant,
  1 or 2 doses:1 on Day 0 and ± 1 on Day 21.
  Other Names: (Monovalent B.1.351 [Beta] variant strain vaccine)
  Arms: Group A- SII B.1.351 Vaccine / Matrix-M1 Adjuvant; Group C- SII B.1.351 Vaccine / Matrix-M1 Adjuvant
Biological: SII B.1.351 — Intramuscular (deltoid) injections of 5 μg SII B.1.351 and 50 μg Matrix-M1 Adjuvant,
  1 or 2 doses:1 on Day 0 and ± 1 on Day 21.
  Other Names: (Monovalent B.1.351 [Beta] variant strain vaccine)
  Arms: Group B- SII B.1.351 Vaccine / Matrix-M1 Adjuvant; Group D - SII B.1.351 Vaccine / Matrix-M1 Adjuvant
Biological: SII Bivalent — Intramuscular (deltoid) injections of 6 μg SII Bivalent and 50 μg Matrix-M1 Adjuvant, 2 doses: 1 on Day 0 and 1 on Day 21.
  Other Names: (Bivalent ancestral and B.1.351 [Beta] variant strain vaccine)
  Arms: Group E -SII Bivalent Vaccine / Matrix-M1 Adjuvant
Biological: SII Bivalent — Intramuscular (deltoid) injections of 10 μg SII Bivalent and 50 μg Matrix-M1 Adjuvant, 2 doses: 1 on Day 0 and 1 on Day 21.
  Other Names: (Bivalent ancestral and B.1.351 [Beta] variant strain vaccine)
  Arms: Group F- SII Bivalent Vaccine / Matrix-M1 Adjuvant
Biological: SII B.1.617.2 — Intramuscular (deltoid) injections of 5 μg SII B.1.617.2 and 50 μg Matrix-M1 Adjuvant,
  1 or 2 doses:1 on Day 0 and ± 1 on Day 21.
  Other Names: (Monovalent B.1.617.2 [Delta] variant strain vaccine)
  Arms: Group G- SII B.1.617.2 Vaccine / Matrix-M1 Adjuvant; Group H- SII B.1.617.2 Vaccine / Matrix-M1 Adjuvant

SUMMARY:
This is a randomized, observer-blinded, Phase 1/2 study with an open-label group to evaluate the safety and immunogenicity of 3 novel SARS-CoV-2 variant vaccine constructs adjuvanted with Matrix-M1 adjuvant. Investigational products will include a monovalent SII SARS-CoV-2 B.1.351 (Beta) variant vaccine (SII B.1.351), a bivalent SII vaccine containing antigen for both the ancestral strain and B.1.351 (Beta) variant of SARS-CoV-2 (SII Bivalent), and a monovalent SII SARS-CoV-2 B.1.617.2 (Delta) variant vaccine (SII B.1.617.2).

ELIGIBILITY:
Inclusion Criteria:

1. Adults 18 to 64 years of age, inclusive, at screening.
2. Willing and able to give informed consent prior to study enrollment and to comply with study procedures.
3. Female participants of childbearing potential (defined as any participant who has experienced menarche and who is NOT surgically sterile [ie, hysterectomy, bilateral tubal ligation, or bilateral oophorectomy] or postmenopausal [defined as amenorrhea at least 12 consecutive months]) must agree to be heterosexually inactive from at least 28 days prior to enrollment and through the end of the study OR agree to consistently use a medically acceptable method of contraception listed below from at least 28 days prior to enrollment and through the end of the study.

   1. Condoms (male or female) with spermicide (if acceptable in country)
   2. Diaphragm with spermicide
   3. Cervical cap with spermicide
   4. Intrauterine device
   5. Oral or patch contraceptives
   6. Norplant®, Depo-Provera®, or other in-country regulatory approved contraceptive method that is designed to protect against pregnancy
   7. Abstinence, as a form of contraception, is acceptable if in line with the participant's lifestyle
4. Is medically stable, as determined by the investigator (based on a review of health status, vital signs [to include body temperature], medical history, and targeted physical examination [to include body weight]). Vital signs must be within medically acceptable ranges prior to the first vaccination.
5. Agrees to not participate in any other SARS-CoV-2 prevention or treatment trials for the duration of the study.

   For previously vaccinated Participants (Groups C, D and H):
6. Documented receipt of 2 doses of the investigational Novavax vaccine with Matrix-M1 adjuvant (NVX-CoV2373) administered approximately 21 days apart or 2 doses of a TGA-authorized/approved COVID-19 vaccine administered at least 60 days prior to first study vaccination.

Exclusion Criteria:

If an individual meets any of the following criteria, he or she is ineligible for this study:

1. History of laboratory-confirmed (by PCR or serology to SARS-CoV-2) COVID-19 infection at any time prior to randomization/enrollment.
2. Previous receipt of any investigational or authorized/approved vaccine, prophylactic or therapeutic agent for the prevention or treatment of SARS-CoV-2 infection, except for previously vaccinated participants.
3. Participation in research involving receipt of investigational products (drug/biologic/device) within 90 days prior to first study vaccination.
4. Received influenza vaccination within 14 days prior to first study vaccination, or any other vaccine within 30 days prior to the first study vaccination.
5. Any known allergies to products contained in the investigational product.
6. Any history of anaphylaxis to any prior vaccine.
7. Autoimmune or immunodeficiency disease/condition (iatrogenic or congenital) requiring ongoing immunomodulatory therapy.
8. Chronic administration (defined as > 14 continuous days) of immunosuppressants, systemic glucocorticoids, or other immune-modifying drugs within 90 days prior to first study vaccination.
9. Received immunoglobulin, blood-derived products, or immunosuppressant drugs within 90 days prior to first study vaccination.
10. Active cancer (malignancy) on therapy within 3 years prior to first study vaccination (with the exception of adequately treated non-melanomatous skin carcinoma or lentigo maligna and uterine cervical carcinoma in situ without evidence of disease, at the discretion of the investigator).
11. Participants who are breastfeeding, pregnant, or who plan to become pregnant prior to the end of study.
12. Suspected or known history of alcohol abuse or drug addiction within 2 years prior to the first study vaccine dose that, in the opinion of the investigator, might interfere with protocol compliance.
13. Any other condition that, in the opinion of the investigator, would pose a health risk to the participant if enrolled or could interfere with evaluation of the study vaccine or interpretation of study results (including neurologic or psychiatric conditions likely to impair the quality of safety reporting).
14. Study team member or immediate family member of any study team member (inclusive of Sponsor, CRO, and study site personnel involved in the conduct or planning of the study).

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2022-02-04 (Estimated); Primary Completion 2022-08 (Estimated); Study Completion 2022-08 (Estimated)

PRIMARY OUTCOMES:
MN50 GMTs to the SARS-CoV-2 B.1.351 (Beta) expressed as GMT | Day 14 and Day 35
  (MN50) geometric mean titers (GMTs) to the SARS-CoV-2 B.1.351 (Beta) variant at Day 14 (one-dose regimen; Groups C and D) and Day 35 (two-dose regimen; Groups A and B);
MN50 GMTs to the SARS-CoV-2 B.1.351 (Beta) expressed as SCRs/SRRs | Day 14 and Day 35
  Seroconversion rates (SCRs) or seroresponse rates (SRRs) (proportion of participants who achieve ≥ 4-fold increase from baseline) in MN50 titer concentrations to the SARS-CoV-2 B.1.351 (Beta) variant following their last vaccination.
MN50 GMTs to the SARS-CoV-2 B.1.617.2 (Delta)expressed as GMT | Day 14 and Day 35
  Neutralizing antibody MN50 GMTs to the SARS-CoV-2 B.1.617.2 (Delta) variant at Day 14 (one-dose regimen; Group H) and Day 35 (two-dose regimen; Group G);
MN50 GMTs to the SARS-CoV-2 B.1.617.2 (Delta)expressed as SCRs/SRRs | Day 14 and Day 35
  SCRs/SRRs (proportion of participants who achieve ≥ 4-fold increase from baseline) in MN50 titer concentrations to the SARS-CoV-2 Delta variant following their last vaccination.
Incidence, duration, and severity of solicited local and systemic adverse events (AEs) | Day 0 to Day 7
  Incidence, duration, and severity of solicited local and systemic adverse events (AEs) for 7 days following each vaccination
Incidence, duration, severity, and relationship of unsolicited AEs through 28 days | Day 0 to Day 28
  Incidence, duration, severity, and relationship of unsolicited AEs through 28 days after the last vaccination
Incidence and relationship of medically attended adverse events (MAAEs), adverse events of special interest (AESIs) (predefined list), and serious adverse events (SAEs) | Day 0 to Day 217
  Incidence and relationship of medically attended adverse events (MAAEs), adverse events of special interest (AESIs) (predefined list), and serious adverse events (SAEs) throughout the study.

SECONDARY OUTCOMES:
MN50 GMTs to the SARS-CoV-2 B.1.351 (Beta) expressed as GMFR in previously vaccinated patients | Day 0 to Day 189
  MN50 GMTs to the SARS-CoV-2 B.1.351 (Beta) variants and to the ancestral SARS-CoV-2 strain at Days 0, 14, and 189 in previously vaccinated individuals
MN50 GMTs to the SARS-CoV-2 B.1.351 (Beta) expressed as GMFR in participants seronegative at baseline | Day 0 to Day 217
  MN50 GMTs to the SARS-CoV-2 B.1.351 (Beta) variants and to the ancestral SARS-CoV-2 strain at Days 0, 21, 35, and 217 in participants seronegative at baseline.
MN50 GMTs to the SARS-CoV-2 B.1.351 (Beta) expressed as SCRs/SRRs in previously vaccinated patients | Day 0 to Day 189
  MN50 GMTs to the SARS-CoV-2 B.1.351 (Beta) variants and to the ancestral SARS-CoV-2 strain at Days 0, 14, and 189 in previously vaccinated individuals
MN50 GMTs to the SARS-CoV-2 B.1.351 (Beta) expressed as SCRs/SRRs in participants seronegative at baseline. | Day 0 to Day 217
  MN50 GMTs to the SARS-CoV-2 B.1.351 (Beta) variants and to the ancestral SARS-CoV-2 strain at Days 0, 21, 35, and 217 in participants seronegative at baseline.
MN50 GMTs to the SARS-CoV-2 B.1.617.2 (Delta) expressed as GMFR in participants seronegative at baseline | Day 0 to Day 217
  MN50 GMTs to the SARS-CoV-2 B.1.617.2 (Delta) variants and to the ancestral SARS-CoV-2 strain at Days 0, 21, 35, and 217 in participants seronegative at baseline.
MN50 GMTs to the SARS-CoV-2 B.1.617.2 (Delta) expressed as GMFR in previously vaccinated participants | Day 0 to Day 189
  MN50 GMTs to the SARS-CoV-2 B.1.617.2 (Delta) variants and to the ancestral SARS-CoV-2 strain at Days 0, 14, and 189 in previously vaccinated individuals
MN50 GMTs to the SARS-CoV-2 B.1.617.2 (Delta)expressed as SCRs/ SRRs in participants seronegative at baseline | Day 0 to Day 217
  MN50 GMTs to the SARS-CoV-2 B.1.617.2 (Delta) variants and to the ancestral SARS-CoV-2 strain at Days 0, 21, 35, and 217 in participants seronegative at baseline.
MN50 GMTs to the SARS-CoV-2 B.1.617.2 (Delta)expressed as SCRs/ SRRs in previously vaccinated participants | Day 0 to Day 189
  MN50 GMTs to the SARS-CoV-2 B.1.617.2 (Delta) variants and to the ancestral SARS-CoV-2 strain at Days 0, 14, and 189 in previously vaccinated individuals
IgG geometric mean concentrations (GMCs) to the SARS-CoV-2 B.1.351 (Beta) expressed as GMFR in previously vaccinated participants | Day 0 to Day 189
  IgG geometric mean concentrations (GMCs) to the SARS-CoV-2 B.1.351 (Beta) variant S proteins and to the ancestral SARS-CoV-2 strain S protein at Days 0, 14, and 189 in previously vaccinated individuals
IgG geometric mean concentrations (GMCs) to the SARS-CoV-2 B.1.351 (Beta) expressed as GMFR in participants seronegative at baseline | Day 0 to Day 217
  IgG geometric mean concentrations (GMCs) to the SARS-CoV-2 B.1.351 (Beta) variant S proteins and to the ancestral SARS-CoV-2 strain S protein at Days 0, 21, 35, and 217 in participants seronegative at baseline.
IgG geometric mean concentrations (GMCs) to the B.1.617.2 (Delta) variant S proteins and to the ancestral SARS-CoV-2 strain S protein in participants seronegative at baseline | Day 0 to Day 217
  IgG geometric mean concentrations (GMCs) to the SARS-CoV-2 B.1.617.2 (Delta) variant S proteins and to the ancestral SARS-CoV-2 strain S protein at Days 0, 21, 35, and 217 in participants seronegative at baseline.
IgG geometric mean concentrations (GMCs) to the B.1.617.2 (Delta) variant S proteins and to the ancestral SARS-CoV-2 strain S protein in previously vaccinated participants | Day 0 to Day 189
  IgG geometric mean concentrations (GMCs) to the SARS-CoV-2 B.1.617.2 (Delta) variant S proteins and to the ancestral SARS-CoV-2 strain S protein at Days 0, 14, and 189 in previously vaccinated individuals
Human Angiotensin-Converting Enzyme 2 (hACE2) receptor binding inhibition assay GMT to the SARS-CoV-2 B.1.351 (Beta) expressed as GMFR in previously vaccinated participants | Day 0 to Day 189
  GMTs to the SARS-CoV-2 B.1.351 (Beta) variant S proteins and to the ancestral SARS-CoV-2 strain S protein at Days 0, 14, and 189 in previously vaccinated individuals
Human Angiotensin-Converting Enzyme 2 (hACE2) receptor binding inhibition assay GMT to the SARS-CoV-2 B.1.351 (Beta) expressed as GMFR in participants seronegative at baseline | Day 0 to Day 217
  GMTs to the SARS-CoV-2 B.1.351 (Beta) variant S proteins and to the ancestral SARS-CoV-2 strain S protein at Days 0, 21, 35, and 217 in participants seronegative at baseline.
Human Angiotensin-Converting Enzyme 2 (hACE2) receptor binding inhibition assay GMT to the SARS-CoV-2 B.1.351 (Beta) expressed as SCRs/SRRs in previously vaccinated participants | Day 0 to Day 189
  GMTs to the SARS-CoV-2 B.1.351 (Beta) variant S proteins and to the ancestral SARS-CoV-2 strain S protein at Days 0, 14, and 189 in previously vaccinated individuals
Human Angiotensin-Converting Enzyme 2 (hACE2) receptor binding inhibition assay GMT to the SARS-CoV-2 B.1.351 (Beta) expressed as SCRs/SRRs in participants seronegative at baseline | Day 0 to Day 217
  GMTs to the SARS-CoV-2 B.1.351 (Beta) variant S proteins and to the ancestral SARS-CoV-2 strain S protein at Days 0, 14, and 189 at Days 0, 21, 35, and 217 in participants seronegative at baseline.
Human Angiotensin-Converting Enzyme 2 (hACE2) receptor binding inhibition assay GMT to the SARS-CoV-2 B.1.617.2 (Delta) expressed as GMFR in participants seronegative at baseline | Day 0 to Day 217
  GMTs to the SARS-CoV-2 B.1.617.2 (Delta) variant S proteins and to the ancestral SARS-CoV-2 strain S protein and at Days 0, 21, 35, and 217 in participants seronegative at baseline.
Human Angiotensin-Converting Enzyme 2 (hACE2) receptor binding inhibition assay GMT to the SARS-CoV-2 B.1.617.2 (Delta) expressed as GMFR in previously vaccinated participants | Day 0 to Day 189
  GMTs to the SARS-CoV-2 B.1.617.2 (Delta) variant S proteins and to the ancestral SARS-CoV-2 strain S protein and at Days 0, 14, and 189 in previously vaccinated individuals
Human Angiotensin-Converting Enzyme 2 (hACE2) receptor binding inhibition assay GMT to the SARS-CoV-2 B.1.617.2 (Delta) expressed as SCRs/SRRs in participants seronegative at baseline | Day 0 to Day 217
  GMTs to the SARS-CoV-2 B.1.617.2 (Delta) variant S proteins and to the ancestral SARS-CoV-2 strain S protein and at Days 0, 21, 35, and 217 in participants seronegative at baseline.
Human Angiotensin-Converting Enzyme 2 (hACE2) receptor binding inhibition assay GMT to the SARS-CoV-2 B.1.617.2 (Delta) expressed as SCRs/SRRs in previously vaccinated participants | Day 0 to Day 189
  GMTs to the SARS-CoV-2 B.1.617.2 (Delta) variant S proteins and to the ancestral SARS-CoV-2 strain S protein and at Days 0, 14, and 189 in previously vaccinated individuals

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Development, Study Director — Novavax
Locations (4):
- Australia (4):
  - Australian Clinical Research Network (ACRN), Maroubra, New South Wales
  - Holdsworth House Medical Practice - Sydney, Sydney, New South Wales
  - University Hospital Geelong-Barwon Health, Geelong, Victoria
  - Emeritus Research, Melbourne, Victoria